CLINICAL TRIAL: NCT00528411
Title: A Multi-centre Randomised, Double-blind, Double-dummy Parallel Group Study of the Onset and Offset of Antiplatelet Effects of Ticagrelor Compared With Clopidogrel and Placebo With Aspirin as Background Therapy in Patients With Stable Coronary Artery Disease (CAD)
Brief Title: A Study of the Onset and Offset of Antiplatelet Effects Comparing Ticagrelor, Clopidogrel, and Placebo With Aspirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5130C00048
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; CAD; heart attack; stable angina; Stable coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina, Stable | interventions — Ticagrelor; Clopidogrel; Capsules; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Aspirin + Placebo
  Interventions: Drug: Aspirin Tablets
- 2 (Active Comparator): Aspirin + clopidogrel
  Interventions: Drug: Clopidogrel (over encapsulated) capsule; Drug: Aspirin Tablets
- 3 (Experimental): Aspirin + Ticagrelor
  Interventions: Drug: Ticagrelor Tablets; Drug: Aspirin Tablets

INTERVENTIONS:
Drug: Ticagrelor Tablets — Oral, 90 mg; 180 mg loading dose followed by 90 mg twice daily (BD)
  Arms: 3
Drug: Clopidogrel (over encapsulated) capsule — Oral 75 mg; 600 mg loading dose followed by 75 mg once daily (ODD)
  Other Names: Plavix; Clopidogrel Bisulfate
  Arms: 2
Drug: Aspirin Tablets — Oral, 75 mg to 100 mg once daily. Aspirin obtained locally by the investigator, according to local practice. The dose remained constant throughout the study.
  Other Names: ASA

SUMMARY:
The purpose of this study is to see how Ticagrelor, a new oral reversible anti-platelet medication, affects platelets. Anti-platelet agents are medications that block the formation of blood clots by preventing the clumping of platelets. Blood clots prevent us from bleeding, but when they form inside the arteries their formation is linked to a risk of medical problems such as heart attack and stroke. This study investigated how long it takes for Ticagrelor to begin working and how long it takes for it to stop working after the last dose of drug. Ticagrelor will be compared to clopidogrel, an established anti-platelet treatment for preventing blood clots, and placebo plus Aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Documented stable Coronary Artery Disease (stable angina, previous MI history, previous history of revascularization);
* Females of child bearing potential must have a negative pregnancy test prior to receiving study drug and be willing to use a hormonal contraceptive in addition to double barrier contraception

Exclusion Criteria:

* History of Acute Coronary Syndromes within 12 months of screening or need for revascularization (angioplasty or Coronary Artery Bypass Graft (CABG))
* History of liver or kidney disease
* Have increased bleeding risk, eg, recent gastrointestinal bleed, uncontrolled high blood pressure, low platelet count, recent major trauma
* History of intolerance or allergy to Aspirin or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Sager, MD, Study Director — AstraZeneca; Paul Gurbel, MD, Principal Investigator — Platelet & Thrombosis Research, LLC
Locations (9):
- United States (8):
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rapid City, South Dakota
  - Research Site, Houston, Texas
- Research Site, Sheffield, United Kingdom

REFERENCES:
- [Derived] Jeong YH, Bliden KP, Antonino MJ, Park KS, Tantry US, Gurbel PA. Usefulness of the VerifyNow P2Y12 assay to evaluate the antiplatelet effects of ticagrelor and clopidogrel therapies. Am Heart J. 2012 Jul;164(1):35-42. doi: 10.1016/j.ahj.2012.03.022. Epub 2012 Jun 13. PMID 22795280
- [Derived] Jeong YH, Bliden KP, Tantry US, Gurbel PA. High on-treatment platelet reactivity assessed by various platelet function tests: is the consensus-defined cut-off of VASP-P platelet reactivity index too low? J Thromb Haemost. 2012 Mar;10(3):487-9. doi: 10.1111/j.1538-7836.2011.04604.x. No abstract available. PMID 22212857
- [Derived] Tantry US, Bliden KP, Wei C, Storey RF, Armstrong M, Butler K, Gurbel PA. First analysis of the relation between CYP2C19 genotype and pharmacodynamics in patients treated with ticagrelor versus clopidogrel: the ONSET/OFFSET and RESPOND genotype studies. Circ Cardiovasc Genet. 2010 Dec;3(6):556-66. doi: 10.1161/CIRCGENETICS.110.958561. Epub 2010 Nov 15. PMID 21079055
- [Derived] Storey RF, Bliden KP, Patil SB, Karunakaran A, Ecob R, Butler K, Teng R, Wei C, Tantry US, Gurbel PA; ONSET/OFFSET Investigators. Incidence of dyspnea and assessment of cardiac and pulmonary function in patients with stable coronary artery disease receiving ticagrelor, clopidogrel, or placebo in the ONSET/OFFSET study. J Am Coll Cardiol. 2010 Jul 13;56(3):185-93. doi: 10.1016/j.jacc.2010.01.062. PMID 20620737
- [Derived] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168

RESULTS

PARTICIPANT FLOW:
Groups:
- Ticagrelor: Ticagrelor 180 mg loading dose followed by 90 mg Twice Daily (bd), plus clopidogrel placebo loading and Once Daily (od) maintenance doses
- Clopidogrel: Clopidogrel 600 mg loading dose followed by 75 mg Twice Daily (od), plus ticagrelor placebo loading and Once Daily (bd) maintenance doses
- Placebo: Ticagrelor 180 mg placebo loading dose followed by 90 mg Twice Daily (bd), plus clopidogrel placebo loading and Once Daily (od) maintenance doses
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Started | 57 | 54 | 12
Completed | 52 | 51 | 11
Not Completed | 5 | 3 | 1
Not completed — Adverse Event | 4 | 0 | 1
Not completed — Incorrect Enrolment | 1 | 1 | 0
Not completed — Severe non-compliance to protocol | 0 | 1 | 0
Not completed — Prior commitment medication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ticagrelor: Ticagrelor 180 mg loading dose followed by 90 mg bd, plus Clopidogrel placebo loading and od maintenance doses
- Clopidogrel: Clopidogrel 600 mg loading dose followed by 75 mg od, plus ticagrelor placebo loading and bd maintenance doses
- Placebo: Ticagrelor 180 mg placebo loading dose followed by 90 mg bd, plus clopidogrel placebo loading and od maintenance doses
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Placebo | Total
Number analyzed (Participants) | 57 | 54 | 12 | 123
Age Continuous [Mean (Standard Deviation); unit: Year] | 62.2 (9.10) | 65.4 (7.98) | 63.9 (8.32) | 63.8 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 2 | 30
  Male | 43 | 40 | 10 | 93

OUTCOME MEASURES:

1. Primary Outcome: Final Extent Inhibition of Platelet Aggregation (IPA) Induced by 20 µM Adenosine Diphosphate (ADP) at 2 Hours After First Dose
Description: IPA(%)=(PAb-PAt)/PAb*100.The unit % is the percentage of difference for baseline versus post baseline value relative to baseline value of platelet aggregation. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: At 2 hours after first dose of study drug
Population: Intent-to-treat analysis set: included patients who were randomised to a treatment group, received at least one dose of study drug, and contributed post baseline data.
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 48 | 49
Percentage | 93.15 [80.4 to 100.0] | 31.05 [10.3 to 56.9]

2. Primary Outcome: Slope of Extent IPA Offset Curve 4 to 72 Hours After Last Dose of Study Drug
Description: IPA(%)=(PAb-PAt)/PAb*100.The unit % is the percentage of difference for baseline versus post baseline value relative to baseline value of platelet aggregation. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition. The unit for the slope of IPA curve is percent/hour.
Time Frame: 4 to 72 Hours after last dose of study drug
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage/Hour
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 54 | 50
Percentage/Hour | -1.037 (0.076) [lower limit 0.076] | -0.482 (0.055) [lower limit 0.055]

3. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 0.5 Hours After First Dose
Description: IPA(%)=(PAb-PAt)/PAb*100. The unit % is the percentage of difference for baseline versus post baseline value relative to baseline value of platelet aggregation. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: 0.5 hours after first dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage | 45.39 [3.0 to 66.4] | 4.71 [0.0 to 14.8]

4. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 1 Hour After First Dose
Description: as for outcome 3
Time Frame: 1 hour after first dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 47 | 47
Percentage | 86.71 [72.6 to 99.4] | 15.83 [0.0 to 32.5]

5. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 4 Hours After First Dose
Description: as for outcome 3
Time Frame: 4 hours after first dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 49 | 48
Percentage | 98.39 [84.2 to 100.0] | 40.87 [16.6 to 69.3]

6. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 8 Hours After First Dose
Description: as for outcome 3
Time Frame: 8 hours after first dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 53 | 47
Percentage | 96.99 [81.1 to 100.0] | 46.90 [20.4 to 80.8]

7. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 24 Hours After First Dose
Description: as for outcome 3
Time Frame: 24 hours after first dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 52 | 46
Percentage | 87.29 [62.9 to 98.4] | 49.64 [17.7 to 76.9]

8. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 0 Hour Before Last Dose
Description: as for outcome 3
Time Frame: 0 hour before last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 44 | 42
Percentage | 74.53 [56.5 to 98.3] | 51.75 [32.8 to 66.4]

9. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 2 Hours After Last Dose
Description: IPA(%)=(PAb-PAt)/PAb*100. The unit % is the percentage of difference for baseline versus post baseline value relative to baseline value. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: 2 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 45 | 43
Percentage | 91.49 [83.0 to 100.0] | 62.96 [35.2 to 78.8]

10. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 4 Hours After Last Dose
Description: as for outcome 3
Time Frame: 4 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 47 | 44
Percentage | 96.10 [80.4 to 100.0] | 61.80 [35.2 to 88.4]

11. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 8 Hours After Last Dose
Description: as for outcome 3
Time Frame: 8 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 47 | 44
Percentage | 88.31 [77.3 to 100.0] | 61.31 [39.0 to 61.31]

12. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 24 Hours After Last Dose
Description: as for outcome 3
Time Frame: 24 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 48 | 45
Percentage | 55.18 [39.1 to 85.4] | 53.91 [35.1 to 73.3]

13. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 48 Hours After Last Dose
Description: as for outcome 3
Time Frame: 48 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 49 | 43
Percentage | 30.94 [14.3 to 51.5] | 45.79 [19.4 to 54.7]

14. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 72 Hours After Last Dose
Description: as for outcome 3
Time Frame: 72 hours after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 49 | 42
Percentage | 11.76 [0.0 to 34.5] | 21.09 [10.2 to 47.6]

15. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 120 Hours - Day 5 After Last Dose
Description: as for outcome 3
Time Frame: 120 hours - Day 5 after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 49 | 41
Percentage | 0.0 [0.0 to 15.2] | 21.15 [0.0 to 34.7]

16. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 168 Hours - Day 7 After Last Dose
Description: IPA(%)=(PAb-PAt)/PAb*100. The unit % is the percentage of difference of baseline versus post baseline value relative to baseline value of platelet aggregation. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: 168 hours - Day 7 after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 47 | 41
Percentage | 0.0 [0.0 to 11.7] | 6.32 [0.0 to 22.4]

17. Secondary Outcome: Final Extent IPA Induced by 20 µM ADP at 240 Hours - Day 10 After Last Dose
Description: as for outcome 3
Time Frame: 240 hours - Day 10 after last dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 48 | 44
Percentage | 1.64 [0.0 to 9.9] | 0.98 [0.0 to 13.8]

18. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is measured by Spirometry, the unit is Liter.
Time Frame: Baseline
Population: Safety analysis set: included all patients who received at least 1 dose of study drug and contribute to the week 1 baseline data.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Liter | 2.79 (0.725) | 2.71 (0.791) | 2.94 (0.654)

19. Secondary Outcome: Cardiopulmonary Parameters at Post 6-week Treatment: FEV1
Description: FEV1 is measured by Spirometry, the unit is Liter.
Time Frame: 6-week post treatment
Population: Safety analysis set: included all patients who received at least 1 dose of study drug and contribute to the week 6 post treatment data.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter | 2.77 (0.712) | 2.74 (0.751) | 2.95 (0.727)

20. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Forced Vital Capacity (FVC)
Description: FVC is measured by Spirometry, the unit is Liter.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Liter | 3.72 (0.903) | 3.73 (1.082) | 4.03 (0.858)

21. Secondary Outcome: Cardiopulmonary Parameters at Post 6-week Treatment: FVC
Description: FVC is measured by Spirometry, the unit is Liter.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter | 3.70 (0.933) | 3.78 (1.029) | 3.98 (0.890)

22. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Ratio of Forced Expiratory Volume in 1 Second Over Forced Vital Capacity (FEV1/FVC Ratio)
Description: FEV1/FVC Ratio is measured by Spirometry, the unit is Ratio.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Ratio | 75.01 (7.049) | 73.04 (6.764) | 73.13 (7.226)

23. Secondary Outcome: Cardiopulmonary Parameters at Post 6-week Treatment: FEV1/FVC Ratio
Description: FEV1/FVC Ratio is measured by Spirometry, the unit is Ratio.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Ratio | 74.71 (5.694) | 72.84 (6.371) | 74.27 (7.836)

24. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Mean Forced Expiratory Flow Between 25% and 75% of the FVC (FEF25-75)
Description: FEF25-75 is measured by Spirometry, the unit is Liter/Second.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter/second
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Liter/second | 2.88 (1.251) | 2.70 (1.208) | 2.50 (1.243)

25. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: FEF25-75
Description: FEF25-75 is measured by Spirometry, the unit is Liter/Second.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter/second
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter/second | 2.77 (1.289) | 2.67 (1.156) | 2.91 (1.375)

26. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Functional Residual Capacity (FRC)
Description: FRC is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 55 | 53 | 12
Liter | 2.79 (0.827) | 2.89 (0.876) | 2.91 (0.679)

27. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: FRC
Description: FRC is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter | 2.73 (0.723) | 2.79 (0.857) | 2.75 (1.000)

28. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Total Lung Capacity (TLC)
Description: TLC is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 55 | 53 | 12
Liter | 5.78 (1.299) | 5.83 (1.401) | 6.10 (1.037)

29. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: TLC
Description: TLC is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter | 5.70 (1.182) | 5.85 (1.396) | 5.96 (1.422)

30. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Residual Volume (RV)
Description: RV is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 55 | 53 | 12
Liter | 1.94 (0.780) | 2.01 (0.643) | 1.91 (0.363)

31. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: RV
Description: RV is measured by Body Box Plethysmography, the unit is Liter.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Liter | 1.88 (0.621) | 1.97 (0.559) | 1.90 (0.751)

32. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Minute Ventilation (VE)
Description: VE is measured by Spirometry and Body Box Plethysmography, the unit is Liter/Minute
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liter/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 55 | 50 | 12
Liter/minute | 12.92 (3.950) | 12.17 (3.552) | 12.06 (4.054)

33. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: VE
Description: VE is measured by Spirometry and Body Box Plethysmography, the unit is Liter/Minute
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 50 | 11
Liter/minute | 13.69 (3.582) | 13.14 (5.515) | 11.45 (3.540)

34. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Respiratory Rate (RR)
Description: RR is measured by Spirometry and Body Box Plethysmography, the unit is Breaths/Minute.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Breaths/minute | 14.79 (2.433) | 14.15 (2.743) | 15.5 (1.977)

35. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: RR
Description: RR is measured by Spirometry and Body Box Plethysmography, the unit is Breaths/Minute.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 52 | 11
Breaths/minute | 15.21 (2.817) | 15.10 (2.303) | 14.91 (0.944)

36. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Tidal Volume (VT)
Description: VT is measured by Body Box Plethysmography, the unit is Liter/Minute.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 55 | 50 | 12
Liters/minute | 0.96 (0.326) | 0.89 (0.322) | 0.89 (0.273)

37. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: VT
Description: VT is measured by Body Box Plethysmography, the unit is Liter/Minute.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 50 | 11
Liters/minute | 0.92 (0.264) | 0.93 (0.393) | 0.83 (0.329)

38. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Single Breath Diffusing Capacity for the Lungs Using Carbon Monoxide (DLCOSB)
Description: DLCOSB is measured by Body Box Plethysmography, the unit is Percent.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Percent | 17.00 (8.673) | 17.29 (10.891) | 15.83 (6.013)

39. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: DLCOSB
Description: DLCOSB is measured by Body Box Plethysmography, the unit is Percent.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 51 | 11
Percent | 16.38 (8.090) | 16.53 (8.286) | 16.09 (7.190)

40. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Ejection Fraction (EF)
Description: EF is measured by Echocardiogram, the unit is Percent. The ejection fraction is defined by: (LV diastolic volume - LV systolic volume)/LV diastolic volume. The unit % is the percentage change of left ventricular diastolic versus systolic volume relative to the diastolic volume. LV is the left ventricle.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 57 | 54 | 12
Percent | 57.96 (9.302) | 61.91 (7.624) | 59.92 (10.013)

41. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: EF
Description: as for outcome 40
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 53 | 52 | 11
Percent | 60.70 (8.430) | 62.38 (7.096) | 60.73 (9.665)

42. Secondary Outcome: Cardiopulmonary Parameters at Baseline: N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP is measured by clinical lab, the unit is pg/mL.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 52 | 53 | 12
pg/ml | 163.34 (184.298) | 185.98 (227.141) | 145.41 (144.522)

43. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: NT-proBNP
Description: NT-proBNP is measured by clinical lab, the unit is pg/mL.
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 43 | 48 | 11
pg/ml | 139.88 (170.347) | 214.43 (313.429) | 140.68 (145.003)

44. Secondary Outcome: Cardiopulmonary Parameters at Baseline: Blood Oxygen Saturation Measured by Pulse Oximetry (SpO2)
Description: SpO2 is measured by pulse oximetry, the unit is Percent. The unit % is the percentage of oxygen attached hemoglobin relative to the total hemoglobin.
Time Frame: Baseline
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 56 | 54 | 12
Percent | 96.59 (1.570) | 96.78 (1.949) | 97.58 (1.240)

45. Secondary Outcome: Cardiopulmonary Parameters Post 6-week Treatment: SpO2
Description: as for outcome 44
Time Frame: 6-week post treatment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Number analyzed (Participants) | 52 | 51 | 9
Percentage | 97.73 (1.239) | 97.35 (1.262) | 98.56 (1.014)

ADVERSE EVENTS:
Arm/Group | Ticagrelor | Clopidogrel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/54 | 0/12
Other Adverse Events (participants affected / at risk) | 36/57 | 22/54 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (N=57) | Clopidogrel (N=54) | Placebo (N=12)
Angina Pectoris (Cardiac disorders) | 3 | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Vessel Puncture Site Haematoma (General disorders) | 3 | 5 | 1
Fatigue (General disorders) | 4 | 2 | 1
Oedema Peripheral (General disorders) | 4 | 2 | 0
Chest Discomfort (General disorders) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 4 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 3 | 0
Electrocardiogram Poor R-Wave Progression (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 6 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 9 | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites.